CLINICAL TRIAL: NCT05044442
Title: Can High Intensity Interval Training Reduce Fear of Hypoglycaemia and Improve Glycaemic Control in People With Type 1 Diabetes?
Brief Title: HIT on Hypoglycaemic Risk in T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: Society for Endocrinology (Other); Royal Liverpool University Hospital (Other Government); University of Birmingham (Other); University of Exeter (Other)
Responsible Party: Principal Investigator, Sam Shepherd, Lecturer/Senior Lecturer, Principle Investigator, Liverpool John Moores University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: SB_T1D_V1
Record Dates: First submitted 2018-06-25; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Type1diabetes
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants will continue with their habitual lifestyle but perform no exercise for 2 weeks
- Moderate intensity continous training (Active Comparator): Participants will complete moderate intensity continous training during a 2 week intervention period
  Interventions: Behavioral: moderate intensity continous training
- high intensity interval training (Experimental): Participants will complete high intensity interval training during a 2 week intervention period
  Interventions: Behavioral: high intensity interval training

INTERVENTIONS:
Behavioral: moderate intensity continous training — Participants will complete 6 sessions of moderate intensity continous training during a 2 week intervention period. Participants will be asked to complete 30 minutes of continuous exercise.
  Arms: Moderate intensity continous training
Behavioral: high intensity interval training — Participants will complete 6 sessions of high intensity interval training during a 2 week intervention period. The programme involves repeated 1 minute bouts of simple on the spot movements interspersed with 1 minute of rest.
  Arms: high intensity interval training

SUMMARY:
There is clear evidence that regular exercise improves wellbeing and reduces the risk of diabetes related complications in people with type 1 diabetes. However, many people with type 1 diabetes do not exercise regularly. The primary reason for this is fear of hypoglycaemia and loss of glycaemic control associated with exercise. This loss of glycaemic control is associated with traditional moderate intensity continous aerobic exercise advocated in the guidelines for exercise in people with type 1 diabetes. Recent work (unpublished) from our lab suggests high intensity interval training (HIT) may reduce the risk of hypoglycaemia in people with type 1 diabetes, however stronger evidence is needed before firm conclusions can be drawn.

Therefore, the aim of this study is to determine the effects of HIT on glycaemic control in people with type 1 diabetes compared to no exercise and traditional moderate intensity continous exercise.

24 people with type 1 diabetes will be recruited to complete a randomised counterbalanced cross over study comparing 3x 2-week interventions periods. During these intervention periods participant will maintain their habitual lifestyle but complete either no exercise (control), traditional moderate intensity continous exercise or high intensity interval training. Throughout the intervention periods participants glycaemic control will be monitored using a flash glucose monitor.

DETAILED DESCRIPTION:
Recruitment 24 people with type 1 diabetes (T1D) will be recruited through local advertising, e.g. within the Liverpool Type 1 Diabetes (LIVT1D) Group.

Protocol The study will use a randomised counterbalanced crossover design, whereby participants will complete 3x 2-week intervention periods; control (no exercise), moderate intensity continous training (MICT) and high intensity interval training (HIT).

Intervention period Participants will complete 3x 2-week intervention periods identical in all respects except for the type of exercise completed.

The day before each intervention period participants will attend the lab at Liverpool John Moores University to have an Abbot Freestyle Libre® flash glucose monitor inserted. To access the data participants will be provide with a "Reader" in "masked" mode, ensuring the participant cannot see the data produced. The Reader will also be used to record time of exercise, insulin doses and blood glucose. Finally, participants will be provided with an activity monitor (Actigraph®) for the duration of the intervention. Participants will also be familiarised to the type of exercise being performed.

In Addition, before the first intervention period participants will also be asked to download MyFitnessPal® to record their daily food intake. An anonymous login email address and password will be given to the participant for access to this App and associated website. A 1ml finger prick blood sample will also be taken on this first visit.

Participants will then complete the 2-week intervention period. During this period participants will be asked to maintain their habitual lifestyle, but only complete the exercise prescribed by the research team (HIT or MICT), or no exercise during the control intervention. Participants will be asked to exercise on day 1, 3, 6, 8, 10 and 13 of the intervention period. Exercise will be completed at any time, but must not be performed following an overnight fast. Participants will be asked to record their blood glucose immediately before and after exercise and 2h post exercise using a finger stick blood sample and automated glucose reader. If participants need to take additional carbohydrates to adjust blood glucose following exercise the investigators will also ask for this to be recorded (what was consumed and time after exercise) using a note in the MyFitnessPal app. Participants will record all insulin doses, time of exercise and food intake for the duration of the intervention period.

Training MICT: Participants will be asked to complete 30 minutes of continuous exercise. Participants will be able to choose any form of exercise (e.g. running or cycling) as long as it is continous in nature. During exercise participants will be asked to maintain a heart rate between 60-70% of their predicted maximum (220-age).

HIT: Participants will be provided with a training guide containing information on the exercises. The programme involves repeated 1 minute bouts of simple on the spot movements interspersed with 1 minute of rest. During the intervals participants will be advised to reach a heart rate of approx. 80% of their predicted maximum heart rate (220-age). The 1 minute interval will be split between 2 consecutive 30 second exercises. The research team have a library of 18 exercises, with 9 suggested exercise pairs. Participants will be advised to complete 6 intervals during each session.

Participants will complete training in a place of their choosing. If requested participants will be able to train in the labs at LJMU.

Participants will be given a polar H7/10 Bluetooth heart rate monitor. Participants will be advised to wear this monitor during all training sessions. The monitor will provide a measure of training intensity and compliance with the suggested heart rate and training programme.

Participants will be asked to download the App PolarBeat to their smartphone. This App will be used to monitor heart rate during the training sessions. In addition, participants will be given a login email address and password for PolarFlow (www.polar.flow.com), a cloud storage site run by Polar for the storage and analysis of heart rate data. All heart rate data measured during training sessions will be uploaded to Polar Flow. This will allow the research team to investigate training intensity achieved during all sessions.

Safety Subjects will be asked to check their blood glucose level to ensure it is safe to exercise. The investigators will use the guidelines that are currently used in a national study of exercise for patients with type 1 diabetes (EXTOD - see attached leaflet). Blood glucose will be checked immediately following exercise and corrected with fast acting carbohydrates if low. The investigators will also advise the subjects to check their glucose level before bed, and if necessary in the early hours of the morning (through setting an alarm clock) if this is required.

Flash Glucose Monitoring Analysis 9 key metrics of glycaemic control will be assessed, reported in 3 time blocks (sleep 00:00-06:00, wake 06:00- 00:00 and 24h 00:00- 00:00): 1) mean glucose, 2) % of time in level 2 hypoglycaemia (<3.0mmol/L), 3) % of time in level 1 hypoglycaemia (3.0-3.9mmol/L), 4) % of time in target range (3.9-10.0mmol/L), 5) % of time in level 1 hyperglycaemia (10.0-13.9mmol/L), 6) % of time in level 2 hyperglycaemia (>13.9mmol/L), 7) glycaemic variability, reported as CV and SD, 8) episodes of hypoglycaemia and hyperglycaemia and 9) area under the curve of episodes of hypoglycaemia and hyperglycaemia.

ELIGIBILITY:
Inclusion Criteria:

* T1D diagnosis more than 6 months ago
* Using a basal bolus insulin regime or insulin pump therapy
* BMI ≤ 32 kg.m-2

Exclusion Criteria:

* Pregnancy (or planning pregnancy)
* Disability preventing participation in an exercise regime
* Angina
* Autonomic neuropathy
* Medication that affects heart rate (this will affect estimation of fitness)
* Major surgery planned within 6 weeks of study
* Uncontrolled blood pressure
* Significant history of hyperglycaemia
* History of severe hypoglycaemia requiring third party assistance within the last 3 months
* Severe non-proliferative and unstable proliferative retinopathy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Severe hypoglycaemia (using continuous glucose monitoring) | Over a 2 week intervention period
  Number of severe hypoglycaemic events (<3mmol/l) during the 2 week intervention period

SECONDARY OUTCOMES:
Mean glucose (using continuous glucose monitoring) | Over a 2 week intervention period
  mean glucose level over 2 week recording period
% of time in level 2 hypoglycaemia (<3.0mmol/L) (using continuous glucose monitoring) | Over a 2 week intervention period
  % of time in level 2 hypoglycaemia (<3.0mmol/L) over 2 week recording period
% of time in level 1 hypoglycaemia (3.0-3.9mmol/L) (using continuous glucose monitoring) | Over a 2 week intervention period
  % of time in level 1 hypoglycaemia (3.0-3.9mmol/L) over 2 week recording period
% of time in target range (3.9-10.0mmol/L) (using continuous glucose monitoring) | Over a 2 week intervention period
  % of time in target range (3.9-10.0mmol/L) over 2 week recording period
% of time in level 1 hyperglycaemia (10.0-13.9mmol/L) (using continuous glucose monitoring) | Over a 2 week intervention period
  % of time in level 1 hyperglycaemia (10.0-13.9mmol/L) over 2 week recording period
% of time in level 2 hyperglycaemia (>13.9mmol/L) (using continuous glucose monitoring) | Over a 2 week intervention period
  % of time in level 2 hyperglycaemia (>13.9mmol/L) over 2 week recording period
glycaemic variability (using continuous glucose monitoring) | 2 weeks
  Standard deviation in glucose concentrations obtained over a 2 week period using a continuous glucose monitoring device.
area under the curve of episodes of hypoglycaemia and hyperglycaemia | Over a 2 week intervention period
  area under the curve of episodes of hypoglycaemia and hyperglycaemia 2 week recording period

CONTACTS AND LOCATIONS:
Locations (1):
- Matthew Cocks, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared outside the research team. Anonymised group data will be presented in research articles and presentations